CLINICAL TRIAL: NCT01898780
Title: Horizontal Mattress vs. Interrupted Suture in Surgical Techniques of Pancreaticojejunostomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Wakayama Medical University (Other)
Responsible Party: Principal Investigator, Hiroki Yamaue, Second Department of Surgery, Wakayama Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOMING
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Patients Who Undergo Pancreatoduodenectomy
MeSH Terms: interventions — Pancreaticojejunostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- horizontal mattress (Experimental): pancreaticojejunostomy with horizontal mattress suture
  Interventions: Procedure: pancreaticojejunostomy with horizontal mattress suture
- interrupted suture (Experimental): pancreaticojejunostomy with interrupted suture
  Interventions: Procedure: pancreaticojejunostomy with interrupted suture

INTERVENTIONS:
Procedure: pancreaticojejunostomy with horizontal mattress suture
  Arms: horizontal mattress
Procedure: pancreaticojejunostomy with interrupted suture
  Arms: interrupted suture

SUMMARY:
The aim of this study is to verify that the frequency of pancreatic fistula (ISGPF grade B and C) in horizontal mattress suture are lower than in interrupted suture during pancreaticojejunostomy in pancreatoduodenectomy by randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

Patients from whom we obtained written informed consent of this study

Exclusion Criteria:

* Patients with severe ischemic cardiac disease
* Patients with severe liver damage
* Patients requiring oxygen administration due to interstitial pneumonia or pulmonary fibrosis
* Patients requiring dialysis treatment due to chronic renal failure
* Patients who are considered as inappropriate by attending physician

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2013-06; Primary Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
The frequency of pancreatic fistula including ISGPF grade B and C | Ninety days after operation

SECONDARY OUTCOMES:
The rates of postoperative complications | Ninety days after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Second Department of Surgery, Wakayama Medical University, Wakayama, Japan

REFERENCES:
- [Derived] Hirono S, Kawai M, Okada KI, Miyazawa M, Kitahata Y, Hayami S, Ueno M, Yamaue H. Modified Blumgart Mattress Suture Versus Conventional Interrupted Suture in Pancreaticojejunostomy During Pancreaticoduodenectomy: Randomized Controlled Trial. Ann Surg. 2019 Feb;269(2):243-251. doi: 10.1097/SLA.0000000000002802. PMID 29697455